CLINICAL TRIAL: NCT01438697
Title: An Internet Intervention for Insomnia: Efficacy and Dissemination
Brief Title: An Interactive Internet Intervention for Adults With Insomnia
Acronym: SHUTi
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Karen Ingersoll, Associate Professor, Department of Psychiatry and NB Sciences, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15704; 1R01MH086758-01A1 (NIH)
Record Dates: First submitted 2011-09-20; First posted 2011-09-22 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Insomnia; Sleep Initiation and Maintenance Disorders
Keywords: sleep; insomnia; internet; CBT
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Internet Intervention (Experimental): Assigned to Sleep Healthy Using the Internet (SHUTi)
  Interventions: Behavioral: Internet Intervention
- Patient Education Website (Active Comparator): Assigned to Patient Insomnia Educational Website
  Interventions: Behavioral: Patient Education Website

INTERVENTIONS:
Behavioral: Internet Intervention — Participants will spend 1-2 hours each week for 9 weeks using the Internet intervention. Users will complete daily sleep diaries as well as interactive tutorials covering the topics of sleep behaviors, sleep thoughts, sleep education, and relapse prevention. As users progress through the program they will receive tailored instructions for how to improve their sleep.
  Other Names: Sleep Healthy Using the Internet (SHUTi)
  Arms: Internet Intervention
Behavioral: Patient Education Website — Participants will be given access to a relevant patient education website. It will contain material addressing the behaviors and symptoms of insomnia.
  Arms: Patient Education Website

SUMMARY:
This study will compare the efficacy of an interactive Internet intervention for adult insomnia (Sleep Healthy Using the Internet; SHUTi) to that of a static educational website to improve sleep, mood related symptoms, perceived health status, and overall quality of life.

DETAILED DESCRIPTION:
Insomnia is defined by complaints of poor sleep, as well as difficulties initiating and/or maintaining sleep more than 3 nights/week for more than 6 months. Insomnia may contribute to daytime fatigue, impaired performance, confused thinking and judgment, and difficulty with work and personal tasks. Cognitive behavioral therapy (CBT) has been found to have significant short- and long-term benefits for people with insomnia. Access to CBT for many people, however, is limited, due to the high cost of treatment and a limited number of trained professionals. Delivering CBT for insomnia via the Internet could help make it more widely available. This study will compare the effectiveness of an online CBT intervention in improving sleep, mood, and quality of life in people with insomnia to that of a static educational website.

Participants in this study will be randomly assigned to receive the online CBT intervention or the static patient education website. The intervention period will last for 9 weeks. During the intervention period, participants assigned to the patient education website will be given content addressing strategies for dealing with insomnia. Those assigned to use the Internet intervention will review interactive, tailored content specific to the user's difficulties. Participants will complete questionnaires and two weeks of daily sleep diaries about their symptoms at four time points - at the beginning of the study, immediately after completing the 9 week program, 6 months later, and 12 months later.

ELIGIBILITY:
Inclusion Criteria:

* Age between 21 and 65 years old.
* Have sleep-onset insomnia and/or sleep maintenance insomnia (>30 minutes for at least 3 nights/week).
* Have insomnia symptoms lasting at least 6 months.
* Have an average total sleep time ≤ 6.5 hours.
* Sleep disturbances (or associated daytime fatigue) cause significant distress or impairment in social, occupational, or other areas of functioning.
* Have regular access to a computer and the Internet.
* Reside in the United States or are US Citizens living outside the United States

Exclusion Criteria:

* Pregnancy
* Report of a physical illness which is deemed active, unstable, degenerative, and/or progressive, such as congestive heart failure, dementia, or acute pain.
* Bipolar disorder as defined by a manic or hypomanic episode or treatment within the past 10 years.
* Severe depression.
* Endorse risk of suicide.
* Endorse alcohol or drug abuse within the past year.
* Presence of another untreated sleep disorder (e.g., sleep apnea, periodic leg movements).
* Have irregular sleep schedules, with usual bedtimes earlier than 8:00pm or later than 2:00am or arising times earlier than 4:00am or later than 10:00am.
* Current psychological treatment for insomnia.
* Initiating psychological treatment within past 3 months.
* Unstable medication regimen (change to schedule or dosage within past 3 months) for a medication regimen thought to impact sleep.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2011-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Primary sleep symptoms: sleep onset latency (SOL), wake after sleep onset (WASO), insomnia severity (ISI) | Baseline, 9 weeks, 6 months, 1 year

SECONDARY OUTCOMES:
Secondary sleep symptoms: sleep efficiency (SE), number of night time awakenings, sleep quality, total sleep time (TST) | Baseline, 9 weeks, 6 months, 1 year
Psychological distress: levels of depression, levels of anxiety, sleep-related cognitions | Baseline, 9 weeks, 6 months, 1 year
Health symptoms: fatigue, quality of life | Baseline, 9 weeks, 6 months, 1 year
Cost effectiveness: program delivery cost, participant resource utilization and costs, quality adjusted life years (QALYs) | 9 weeks, 6 months, 1 year
Intervention Evaluation: perceived utility, perceived impact, intervention adherence, intervention use | 9 weeks, 6 months, 1 year
Exploratory Outcome Measures: health care access, coverage and utilization | Baseline, 9 weeks, 6 months, 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Karen Ingersoll, PhD, Principal Investigator — University Of Virginia Behavioral Health & Technology; Lee M Ritterband, PhD, Study Director — University of Virginia Behavioral Health & Technology
Locations (1):
- University Of Virginia Health System, Department of Psychiatry and Neurobehavioral Sciences, Division of Behavioral Health and Technology, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Thorndike FP, Ritterband LM, Gonder-Frederick LA, Lord HR, Ingersoll KS, Morin CM. A randomized controlled trial of an internet intervention for adults with insomnia: effects on comorbid psychological and fatigue symptoms. J Clin Psychol. 2013 Oct;69(10):1078-93. doi: 10.1002/jclp.22032. Epub 2013 Aug 28. PMID 24014057
- [Result] Quigg M, Gharai S, Ruland J, Schroeder C, Hodges M, Ingersoll KS, Thorndike FP, Yan G, Ritterband LM. Insomnia in epilepsy is associated with continuing seizures and worse quality of life. Epilepsy Res. 2016 May;122:91-6. doi: 10.1016/j.eplepsyres.2016.02.014. Epub 2016 Mar 2. PMID 26994361
- [Result] Ritterband LM, Thorndike FP, Ingersoll KS, Lord HR, Gonder-Frederick L, Frederick C, Quigg MS, Cohn WF, Morin CM. Effect of a Web-Based Cognitive Behavior Therapy for Insomnia Intervention With 1-Year Follow-up: A Randomized Clinical Trial. JAMA Psychiatry. 2017 Jan 1;74(1):68-75. doi: 10.1001/jamapsychiatry.2016.3249. PMID 27902836
- See also: Sleep Health Using the Internet intervention site — http://www.shuti.org
- See also: University of Virginia Behavioral Health & Technology research lab — http://bht.virginia.edu